CLINICAL TRIAL: NCT06635746
Title: Phase I, Open Label, Dose-Escalation Study for Maximum Tolerated Vinpocetine Dose in Healthy Volunteers
Brief Title: Dose Escalation Study of Vinpocetine in Healthy Volunteers
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Kimford Jay Meador, Professor of Neurology, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Protocol: 77615; R61AA031291 (NIH)
Record Dates: First submitted 2024-10-08; First posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Fetal Alcohol Spectrum Disorders
Keywords: Cognition; Vinpocetine
MeSH Terms: conditions — Fetal Alcohol Spectrum Disorders | interventions — vinpocetine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Vinpocetine (Experimental): Participants will take increasing, single doses of vinpocetine.
  Interventions: Drug: Vinpocetine

INTERVENTIONS:
Drug: Vinpocetine — Increasing doses of vinpocetine to assess tolerability.

SUMMARY:
The objective of this study is to determine whether vinpocetine is safe when taken at higher doses.

DETAILED DESCRIPTION:
The planned study seeks to provide preliminary data to assess the benefits and safety for vinpocetine to address cognitive problems in two groups of patients. One group are patients with epilepsy in whom cognitive problems are common, but there is currently no specific treatment available. Vinpocetine has been shown to improve memory in animals and also has anticonvulsant activity. The other group are people who suffer cognitive/behavioral problems from fetal exposure to alcohol or anticonvulsant drugs. In animals, vinpocetine has been shown to mitigate these deficits. We propose to extend our prior preliminary studies by conducting a Phase I study in healthy volunteers, a Phase I study in adolescents with cognitive impairments from fetal alcohol exposure, then Phase II studies in patients with epilepsy and in adolescents/adults with cognitive impairments from fetal alcohol or antiseizure medication (e.g., valproate) exposure. The proposed investigations are guided by prior PK and PD studies in animals and humans. They are designed to provide data on the dosages needed to provide levels comparable to effective animal studies and provide data on the potential efficacy and safety of vinpocetine in improving cognition in order to direct more definitive randomized trials in the future.

Specific Aim: To determine the maximum tolerated oral dose of vinpocetine in healthy adult volunteers and develop data on pharmacokinetic response curve for vinpocetine effects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults 18-40 years old.
2. Proficient English.
3. Use of appropriate contraception if woman of childbearing potential.

Exclusion Criteria:

1. Major medical disease (e.g., epilepsy, diabetes, heart disease, active cancer, depression).
2. Those who score >18 overall on the BDI-II or >0 for item #9 (suicidal thoughts) at screening.
3. Use of centrally active medications.
4. History of allergy to vinpocetine.
5. IQ<80.
6. BMI≥30.
7. Pregnancy or lactation.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | Approximately weekly treatments across ~4-6 visits per participant.
  Safety Outcome

IPD SHARING:
Plan to Share IPD: Undecided
Pending information from funding agency.